CLINICAL TRIAL: NCT02791971
Title: SpeakOut: Empowering Teen to Teen Social Communication About Highly Effective Contraception (Also Known As: The Share Health Study: Teen Social Connections and Health)
Brief Title: The Share Health Study: Teen Social Connections and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP2AH000045-01-01
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Contraception
Keywords: Contraception; Birth control; Social communication; Adolescent; Social network; Health education; Reproductive health
MeSH Terms: conditions — Communication; Health Education | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SpeakOut Intervention (Experimental): Primary participants will be randomized to this arm or the Alcohol Control Arm at the time of enrollment. Secondary participants will be assigned to this arm if the primary participant whom initially told them about the study is in this arm. Primary participants in this arm will receive the SpeakOut intervention on the day of enrollment, and will complete surveys on their contraceptive knowledge, attitudes, behaviors, and social communication at baseline, three months, and nine months. Secondary participants in this arm will complete similar surveys at baseline, three months, and nine months.
  Note: Secondary participants will not receive intervention, but will be assessed on outcomes that may have been affected as a result of social communication with primary participants.
  Interventions: Behavioral: SpeakOut
- Alcohol Control Intervention (Active Comparator): Primary participants will be randomized to this arm or the SpeakOut Intervention Arm at the time of enrollment. Secondary participants will be assigned to this arm if the primary participant whom initially told them about the study is in this arm. Primary participants in this arm will receive the Alcohol Control Intervention on the day of enrollment, and will complete surveys on their contraceptive knowledge, attitudes, behaviors, and social communication at baseline, three months, and nine months. Secondary participants in this arm will complete similar surveys at baseline, three months, and nine months.
  Note: Secondary participants will receive an intervention, but will be assessed on outcomes that may have been affected as a result of social communication with primary participants.
  Interventions: Behavioral: Alcohol Control Intervention

INTERVENTIONS:
Behavioral: SpeakOut — SpeakOut aims to increase social communication about IUDs and implants between adolescent IUD and implant users and their peers. SpeakOut has four components:
  * Coaching session. Research staff will deliver a script to encourage recipients to share information about their contraceptive method with peers.
  * Printed materials for recipients to keep and/or share with friends.
  * Websites with information and resources. Staff will refer recipients to a website, either SpeakOutIUD.org or SpeakOutImplant.org, which contain information about their method.
  * Text messages with information about recipients' method and about how to share their experience. Recipients will be given the opportunity to sign up for text messages that will be sent for 8 weeks following receipt of SpeakOut in clinic.
  Arms: SpeakOut Intervention
Behavioral: Alcohol Control Intervention — The active comparator intervention is an alcohol assessment and education intervention using an SBIRT (Screening, Brief Intervention, and Referral to Treatment) framework. SBIRT is an evidence-based practice model aimed at preventing problematic use and identifying potential abuse and dependency issues. Research staff will ask two screening questions developed by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) and the American Academy of Pediatrics to screen for adolescents potentially at risk. Using a script based on tenets of motivational interviewing to assess alcohol related consequences, the research staff will guide teens in identifying personally relevant motivators for healthier behaviors, assess readiness to change, and offer educational materials and referrals.
  Other Names: Partywise, Partysafe
  Arms: Alcohol Control Intervention

SUMMARY:
The purpose of this study is to determine whether delivery of SpeakOut, a behavioral intervention to increase social communication about long-acting reversible contraceptive (LARC) methods among adolescents, is associated with increased uptake of LARC methods among the social contacts of SpeakOut recipients.

The investigators will conduct a cluster randomized controlled trial of SpeakOut with adolescent LARC users and their female peers. Over three years, SpeakOut will be implemented in eight partner clinics. IUD and implant users aged 15 to 19 who attend appointments at participating clinics will be invited to enroll in the evaluation study as "primary" participants and receive either SpeakOut or a control intervention about alcohol use. The social contacts of primary participants will be asked to enroll in the study as "secondary" participants. The study's primary outcome will be the proportion of sexually-active secondary participants who initiate use of a LARC method within 9 months of study enrollment.

DETAILED DESCRIPTION:
Teen pregnancy results from sexually active adolescents' under-use of effective contraception. The most effective reversible methods - intrauterine devices (IUDs) and subdermal contraceptive implants, collectively referred to as long-acting reversible contraception (LARC) - have low rates of use among adolescents. Social networks are important influences on teen contraceptive knowledge and use. Encouraging social communication to increase knowledge and acceptability of LARC among female adolescents can increase use of these methods.

The Share Health Study is a cluster randomized control trial, randomized at the primary participant level. Primary participants will be randomized to receive either SpeakOut or a control intervention about alcohol use immediately before intervention delivery on the day of their clinic appointment. A cluster consists of primary participants and the secondary participants recruited to the study via a specialized snowball sampling procedure carried out with the assistance of the primary participant, described below.

The design of SpeakOut was initially motivated by a qualitative study performed by Dr. Dehlendorf's team that found that adolescent IUD users report that a lack of social communication about this method is a barrier to IUD use. Dr. Dehlendorf's team then performed further qualitative work designed to understand the transmission of information about contraception within social networks, with the goal of informing a social-network-based intervention. The investigators confirmed that social communication is an influential factor in contraceptive decision making, and that it is considered particularly important to speak to individuals who have personal experience with specific methods. However, participants reported often hearing negative information about these methods, particularly IUDs, through their social network.

Primary participant procedures

* Partner clinic and affiliate staff will notify research staff of appointment times for female patients aged 15 to 19 who are using or are planning to initiate use of LARC.
* Research staff will approach patients in the clinic waiting room or other clinic area before or after their appointment with approval of clinic staff and invite them to learn more about the study in a private room and be screened for eligibility.
* After being screened and providing written consent, each primary participant will complete a baseline survey collecting demographic information and asking about contraceptive knowledge, attitudes, use, and social communication as well as drug and alcohol behaviors, and will provide a list of first names of female social contacts age 15 to 19 with whom they feel comfortable talking about personal issues. These people will be potential secondary participants for the study. Research staff will ask that in the two weeks after enrollment, primary participants ask potential secondary participants if they are interested in being contacted by research staff, and if they are, to share their contact information with research staff.
* Participants will be randomized to receive either SpeakOut or a control intervention and receive the assigned intervention immediately after randomization.
* Research staff will randomize and deliver the assigned intervention before or after the clinic visit, depending on clinic flow.
* Once randomized, research staff will deliver either SpeakOut or the control intervention to the participant. Each delivery session lasts about 15 minutes, and sessions will be audio-recorded and observed for quality and fidelity measurement by UC Davis staff. As indicated the consent form for primary participants, primary participants may verbally indicate that they do not wish for the session to be recorded, and research staff will not record their session.
* Research staff will complete a fidelity checklist indicating which intervention components the primary participant received.
* Research staff will send primary participants an email and/or text reminder about secondary participant recruitment one week after their enrollment.
* In the period two to four weeks following primary participant enrollment, research staff will contact primary participants so that primary participants may share with research staff which potential secondary participants from their lists are willing to be contacted, as well as potential secondary participants contact information including phone number and/or email.
* Three months after enrollment, research staff will contact primary participants by phone call, text, and/or e-mail and ask them to complete the first follow-up survey over the phone or online. The survey will include questions about contraceptive knowledge, attitudes, and use as well as drug and alcohol behaviors. Research staff will attempt to reach primary participants for up to one month following the 3-month post-enrollment date.
* Nine months after enrollment, research staff will contact primary participants by phone call, text, and/or e-mail and ask them to complete the second follow-up survey over the phone or by-email. The survey will include questions about contraceptive knowledge, attitudes, and use as well as drug and alcohol behaviors. Research staff will attempt to reach primary participants for up to one month following the 9-month post-enrollment date.

In addition to the above procedures, research staff at UC Davis will seek to obtain publically available claims data related to primary participants' reproductive health care over the 9-month study period. If available, Family PACT (Family Planning Access, Care, and Treatment) and Medi-Cal data will be obtained on pregnancy and removal of IUD or implant over the 9-month study period. This data will validate primary participant self-report of pregnancy and method removal at follow-up, or substitute for missing follow-up data. The California Department of Health Care Services (DHCS) has a standardized application process for the evaluation, review and potential approval of requests for protected data for research purposes. To obtain Family PACT and Medi-Cal administrative data from DHCS, researchers must submit an application for approval from the Data and Research Committee (DRC), which oversees DHCS' data request evaluation process, and from the Committee for the Protection of Human Subjects under the California Health and Human Services Agency (CHHSA). The DRC assesses the appropriateness of requests for protected data, assigns a priority status to each request, and recommends potential approval/denial action to DHCS Executive management. As a part of accessing DHCS data, researchers are required to provide a presentation of their findings to DHCS staff. In addition, requests can only be approved if they have a clear and strong argument that the proposed research request will result in information that benefits the Medi-Cal program (Section 1902(a) of the federal Social Security Act (42 U.S.C. 1396a(7)). Linkages to external data sources must be performed by DHCS staff, therefore SpeakOut will need to provide identifiable participant data to DHCS in order to obtain linked administrative data from participants' claims history.

Information about the above process is included in the primary participant consent form, and primary participants may verbally inform the consenting researcher that they opt out of having their data accessed.

Secondary participant procedures

* Potential secondary participants, identified by primary participants at baseline, will initially be approached by the primary participant who listed them. Primary participants will ask for potential secondary participants' permission to be contacted by research staff. Primary participants will report permission to research staff, who will then obtain secondary contact information from primary participants and contact potential secondary participants by phone call, text, and/or e-mail to ask if they would like to screen for eligibility as a secondary participant over the phone. Research staff will attempt to reach potential secondary participants for up to four weeks following primary participant enrollment.
* Eligibility screening will take place over the phone and verbal consent will be obtained.
* Secondary participants will complete a baseline survey collecting demographic information and asking about contraceptive knowledge, attitudes, use, and social communication, as well as drug and alcohol behaviors.
* Three months after enrollment of their primary participant, research staff will contact secondary participants by phone call, text, and/or e-mail and ask them to complete the first follow-up survey over the phone or by-email. The survey will include questions about contraceptive knowledge, attitudes, use, and social communication as well as drug and alcohol behaviors. Research staff will attempt to reach primary participants for up to one month following the 3-month post-enrollment date.
* Nine months after enrollment of their primary participant, research staff will contact secondary participants by phone call, text, and/or e-mail and ask them to complete the second follow-up survey over the phone or by-email. The survey will include questions about contraceptive knowledge, attitudes, and use as well as drug and alcohol behaviors. Research staff will attempt to reach primary participants for up to one month following the 9-month post-enrollment date.

Please note that our sample size of 2500 is based on an estimate of cluster sizes of 4 secondary participants per 1 primary participant. As per our initial grant application, "During the course of the study, the distribution of initial cluster sizes (i.e. enrolled eligible secondary participants per primary participant) will be monitored for gross departures from our planning assumptions. In case of discrepancies, the targeted enrollment will be adjusted to achieve the necessary effective sample size. To preserve the integrity of the trial, this monitoring will only concern enrollment information, not study outcomes."

ELIGIBILITY:
Primary Participant Inclusion Criteria:

* Able to speak and read English or Spanish easily
* Uses an IUD or implant for birth control, or will get one of these methods inserted at an appointment on the day of enrollment
* Is comfortable with close friend knowing that they use an IUD or implant
* Can think of at least one friend or family member they would be comfortable asking to join a study about health topics like birth control and alcohol use

Primary Participant Exclusion Criteria:

* Previous enrollment as a primary or secondary participant in the study
* Pregnant at baseline
* Plan to get their IUD or implant removed at their visit and not replacing it with another LARC

Secondary Participant Inclusion Criteria:

* Able to speak and read English or Spanish easily
* Was listed as a social contact by a primary participant at enrollment, and can name that primary participant at screening
* Lives in California

Secondary Participant Exclusion Criteria:

* Pregnant at baseline
* Previous enrollment as a primary or secondary participant in the study

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 207 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Initiation of a LARC method among secondary participants | 3 months and 9 months post-enrollment
  Self-reported measure of current contraceptive use in secondary participants not using IUD or implant at baseline. Will be examined among sexually active secondary participants, as well as all secondary participants regardless of sexual activity.

SECONDARY OUTCOMES:
Initiation of cluster primary participant's LARC method among secondary participants | 3 months and 9 months post-enrollment
  Self-reported measure of current contraceptive use in secondary participants not using IUD or implant at baseline. Will be examined among sexually active secondary participants, as well as all secondary participants regardless of sexual activity. Outcome will also be examined separately by LARC method, i.e. implant initiation among all secondary participants not using an implant at baseline (even if they used an IUD at baseline) if the primary participant was an implant user, as well as IUD initiation among all secondary participants not using an IUD at baseline (even if they used an implant) if the primary participant was an IUD user.
Positive social communication about LARC method between primary and secondary participants | 3 months and 9 months post-enrollment
  Self-reported measures of discussion about contraceptive methods with primary participant, in secondary participant follow-up surveys, and 5-point likert scale measures of agreement/disagreement with statements of positive and negative content of discussion.
Knowledge of cluster primary participant's LARC method among secondary participants | 3 months and 9 months post-enrollment
  Secondary participants' accurate knowledge of features of their cluster primary participant's LARC method. In baseline and follow-up surveys, secondary participants will be asked to report whether or not they have ever heard of the method. If they have heard of the method in follow-up surveys, they will be asked to report on a 4-point Likert scale their self-perceived knowledge of the method. They will also be asked to answer a set of true/false/don't know knowledge items on the method's features derived from the Guttmacher Institute's Survey of Young Adults ("Fogzone" survey) and National Survey of Reproductive and Contraceptive Knowledge, as well as an item on the relative effectiveness of the method in relation to birth control pills.
Positive attitudes towards cluster primary participant's LARC method among secondary participants | 3 months and 9 months post-enrollment
  Self-reported global attitudinal scales of contraceptive methods in secondary participant baseline and follow-up surveys, scored from 0-10.
Diagnosis of sexually transmitted infection among secondary participants | 3 months and 9 months post-enrollment
  Diagnosis of a sexually transmitted infection (chlamydia, gonorrhea, trichomoniasis [or trich], or other). Measured via self-report in secondary participant follow-up surveys (binary yes/no measure of diagnosis, and measure regarding which STI they were diagnosed with).
Condom use at last sexual intercourse among sexually active secondary participants | 3 months and 9 months post-enrollment
  Self-reported in secondary participant baseline and follow-up surveys with standardized question from the Office of Adolescent Health in the Department of Health and Human Services.
Initiation of sexual activity among secondary participants | 3 months and 9 months post-enrollment
  Self-reported measure of ever having had sexual intercourse (standardized OAH measure) in secondary participant baseline and follow-up surveys among those who had not had sexual intercourse prior to enrollment.
Pregnancy among secondary participants | 3 months and 9 months post-enrollment
  Self-reported measure of interval pregnancy (standardized OAH measure) in secondary participant follow-up surveys.
Continuation of LARC method among primary participants | 3 months and 9 months post-enrollment
  Self-reported measure of current contraceptive method use in primary participant follow-up surveys. Also assessed using claims data.
Initiation of social communication about LARC method among primary participants | 3 months and 9 months post-enrollment
  Primary participants' report of social communication about their LARC method, as well as the number of social contacts they talked to about their LARC method. Self-reported in measures assessing discussion about contraceptive methods with people they know generally and social contacts they listed at baseline specifically in primary participant surveys.
Knowledge of LARC method among primary participants | 3 months and 9 months post-enrollment
  Primary participants' accurate knowledge of their chosen LARC method. In follow-up surveys, they will be asked to report on a 4-point Likert scale their self-perceived knowledge of the method. They will also be asked to answer a set of true/false/don't know knowledge items on the method's features derived from the Guttmacher Institute's Survey of Young Adults ("Fogzone" survey) and National Survey of Reproductive and Contraceptive Knowledge, as well as an item on the relative effectiveness of the method in relation to birth control pills.
Positive attitudes towards LARC method among primary participants | 3 months and 9 months post-enrollment
  Self-reported global attitudinal scales in primary participant baseline and follow-up surveys, scored from 0-10.
Pregnancy among primary participants | 3 months and 9 months post-enrollment
  Self-reported measure of interval pregnancy (standardized OAH measure) in primary participant follow-up surveys.
Risk of unintended pregnancy | 3 months and 9 months post-enrollment
  Participants' risky sexual activity, defined as reporting sex without a contraceptive method in the past 3 months. Self-reported in primary and secondary participants' baseline and follow-up surveys. Will include sub-analysis of both primary and secondary participants.
Alcohol use | 3 months and 9 months post-enrollment
  Participants' days of alcohol use as reported in surveys, measured via self-report in measure derived from the Youth Risk Behavior Survey.
Knowledge of binge-drinking behaviors | 3 months and 9 months post-enrollment
  Participants' knowledge of what constitutes binge drinking, including sex differences in binge drinking. Knowledge measures on follow-up surveys will are derived from the youth Risk Behavior survey.
Diagnosis of an STI among primary participants | 3 months and 9 months post-enrollment
  Diagnosis of a sexually transmitted infection (chlamydia, gonorrhea, trichomoniasis [or trich], or other). Measured via self-report in primary participant follow-up surveys (binary yes/no measure of diagnosis, and measure regarding which STI they were diagnosed with). Also assessed via claims data.
Acceptability of SpeakOut | 9 months
  Measured using items developed by the researchers to understand participants' experience with and opinion of different intervention components of SpeakOut.. Will be examined among both primary and secondary participants.
Acceptability of PartyWise [control intervention] | 9 months
  Measured using items developed by the researchers to understand participants' experience with and opinion of different intervention components of Party Wise. Will be examined among both primary and secondary participants.

OTHER OUTCOMES:
Contraceptive attitudes | 3 months and 9 months post-enrollment
  Participants' attitudes towards various contraceptive methods, reported in global attitudinal scales in surveys, scored from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dehlendorf, MD MAS, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, Davis, California
  - University of Southern California Keck School of Medicine, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided